CLINICAL TRIAL: NCT03533647
Title: A Longitudinal Study on the Development and Pathological Changes Among Children and Adolescents With High Myopia in China
Brief Title: Development and Pathological Changes of High Myopia Among Children and Adolescents in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Clinical Professor,director of Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: SYSU-OPH-003
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: High Myopia
Keywords: high myopia; ocular biometric parameters; adolescent; children
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- entire cohort (observational): none (observational study)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — none (observational study)

SUMMARY:
The study aims to observe the relationship between the changes of ocular structure parameters and pathological changes among children and adolescents with high myopia. Environmental factors and family history will also be collected to explore their impacts on high myopia progression.

DETAILED DESCRIPTION:
This study aims to observe children and adolescents with high myopia for 3 years, and to collect data of ocular pathological changes, family history and environmental factors so as to understand the natural course and internal laws of the development of high myopia.

ELIGIBILITY:
Inclusion Criteria:

* 9 to 18 years old school students in Guangzhou, with either eye had myopia equal or greater than 6.0D
* Or 6 to 8 years old school students in Guangzhou, with either eye had myopia equal or greater than 3.0D
* Written informed consent for study participation
* Be willing to cooperate with the relevant ophthalmological examination and complete the questionnaire.

Exclusion Criteria:

* None school students in Guangzhou
* Other contraindications
* A history of allergy to tropicamide or topical anesthetics
* Missing ability to give informed consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 6 to 18 years old school students in Guangzhou. Age between 9-18 years old with either eye had myopia equal or greater than 6.0D ,age between 6-8 years old with either eye had myopia equal or greater than 3.0D
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2021-05-13 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
To observe the relationship between the changes of ocular structure parameters and pathological changes among children with high myopia. | examine every 12 months, follow up 3 years
  examine the ocular pathological changes

SECONDARY OUTCOMES:
To explore the impact of environmental factors and genetic factors on the progression among children and adolescents with high myopia | examine every 12 months, follow up 3 years
  axial length, refractive error changes, environmental factors, family history, exercise time, eye care habits, form of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi LIU, MD,PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yet-san University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Lin LL, Shih YF, Hsiao CK, Chen CJ. Prevalence of myopia in Taiwanese schoolchildren: 1983 to 2000. Ann Acad Med Singap. 2004 Jan;33(1):27-33. PMID 15008558
- [Background] Sun J, Zhou J, Zhao P, Lian J, Zhu H, Zhou Y, Sun Y, Wang Y, Zhao L, Wei Y, Wang L, Cun B, Ge S, Fan X. High prevalence of myopia and high myopia in 5060 Chinese university students in Shanghai. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7504-9. doi: 10.1167/iovs.11-8343. PMID 23060137
- See also: sample size reference — http://www.raosoft.com/samplesize.html